CLINICAL TRIAL: NCT01009450
Title: Clipless Laparoscopic Cholecystectomy Using Harmonic Scalpel in Cirrhotic Patients a Prospective Randomized Study
Acronym: CLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Mansoura University, Mansoura University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: clipless cholecystectomy
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2009-11-06 (Estimated); Status verified 2009-11

CONDITIONS: Gall Bladder Stone in Cirrhotics
Keywords: cirrhotic liver, gall bladder stone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LC was done using traditional method (Active Comparator): LC was done using traditional method by dissection of calot's triangle and clipping of both cystic duct and artery by metal clips. Then dissection of gall bladder from its bed by hook using electrocautery technique. Finally we insert abdominal drain in Morrison pouch.
  Interventions: Procedure: LC was done using traditional method
- LC was done using harmonic ACE (Active Comparator): LC was done using harmonic ACE (Ethicon Endo-Surgery) by dissection of calot's and then occlusion of both cystic duct and artery using harmonic ACE. For closure of and division of cystic pedicle we set the instrument at a power 2 i.e. more coagulation. And when dissecting the gall bladder from the bed we set it to the level 5 i.e. more cutting power. And control of any bleeding from the bed using the active blade of harmonic ACE. Finally we insert abdominal drain in Morrison pouch.
  Interventions: Procedure: LC was done using harmonic ACE

INTERVENTIONS:
Procedure: LC was done using traditional method — LC was done using traditional method by dissection of calot's triangle and clipping of both cystic duct and artery by metal clips. Then dissection of gall bladder from its bed by hook using electrocautery technique. Finally we insert abdominal drain in Morrison pouch.
  Other Names: traditional laparoscopic cholecystectomy
  Arms: LC was done using traditional method
Procedure: LC was done using harmonic ACE — LC was done using harmonic ACE (Ethicon Endo-Surgery) by dissection of calot's and then occlusion of both cystic duct and artery using harmonic ACE. For closure of and division of cystic pedicle we set the instrument at a power 2 i.e. more coagulation. And when dissecting the gall bladder from the bed we set it to the level 5 i.e. more cutting power. And control of any bleeding from the bed using the active blade of harmonic ACE. Finally we insert abdominal drain in Morrison pouch.
  Other Names: clipless laparoscopic cholecystectomy
  Arms: LC was done using harmonic ACE

SUMMARY:
This study included group (A) (60 patients with liver cirrhosis and complaining of gall stone) in whom LC was done using traditional method (TM) by clipping both cystic duct and artery and dissection of gall bladder from liver bed by diathermy, and group (B) (60 patients with liver cirrhosis and complaining of gall stone) LC was done using harmonic scalpel (HS) closure and division of both cystic duct, artery and dissection of gall bladder from liver bed by harmonic scalpel. The Intraoperative and postoperative parameters were collected included duration of operation, postoperative pain, and complications.

DETAILED DESCRIPTION:
Under general anesthesia, and same antibiotics (3rd generation cephalosporin) Surgery was performed using conventional four ports umbilical port, port below xiphoid and two ports below right costal margin. Pneumoperitoneum at pressure 12 mmHg was used.

In group (A) LC was done using traditional method by dissection of calot's triangle and clipping of both cystic duct and artery by metal clips. Then dissection of gall bladder from its bed by hook using electrocautery technique. Finally we insert abdominal drain in Morrison pouch.

In group (B) LC was done using harmonic ACE (Ethicon Endo-Surgery) by dissection of calot's and then occlusion of both cystic duct and artery using harmonic ACE. For closure of and division of cystic pedicle we set the instrument at a power 2 i.e. more coagulation. And when dissecting the gall bladder from the bed we set it to the level 5 i.e. more cutting power. And control of any bleeding from the bed using the active blade of harmonic ACE. Finally we insert abdominal drain in Morrison pouch.

The Intraoperative parameter observed included duration of the operation, bile escape and volume of blood loss were recorded The patients started oral feeding 8 h postoperatively; abdominal ultrasound was done for all patients in both groups on day of discharge to show any collection or free fluid in the abdomen. The patients were usually discharged after removal of drain, and when the patient surgically free.

Postoperative pain was evaluated at 12 h, 24h, 48, 1 w after operation using a visual analog scale (VAS)

ELIGIBILITY:
Inclusion Criteria:

* patients with liver cirrhosis with symptomatic gall bladder stone

Exclusion Criteria:

* patients above 80 years old,
* patients with history of upper laparotomy,
* patients with common bile duct stones
* and pregnant females.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
time of operation,pain,and bleeding | 14 days postoperative

SECONDARY OUTCOMES:
complications | 30 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: ayman el nakeeb, MD, Principal Investigator — Mansoura University Hospital
Locations (1):
- Ayman El Nakeeb, Al Mansurah, Mansoura, Egypt

REFERENCES:
- [Result] Kandil T, El Nakeeb A, El Hefnawy E. Comparative study between clipless laparoscopic cholecystectomy by harmonic scalpel versus conventional method: a prospective randomized study. J Gastrointest Surg. 2010 Feb;14(2):323-8. doi: 10.1007/s11605-009-1039-8. Epub 2009 Oct 31. PMID 19882194
- [Result] El-Awadi S, El-Nakeeb A, Youssef T, Fikry A, Abd El-Hamed TM, Ghazy H, Foda E, Farid M. Laparoscopic versus open cholecystectomy in cirrhotic patients: a prospective randomized study. Int J Surg. 2009 Feb;7(1):66-9. doi: 10.1016/j.ijsu.2008.10.013. Epub 2008 Oct 26. PMID 19028148
- [Result] Ji W, Li LT, Wang ZM, Quan ZF, Chen XR, Li JS. A randomized controlled trial of laparoscopic versus open cholecystectomy in patients with cirrhotic portal hypertension. World J Gastroenterol. 2005 Apr 28;11(16):2513-7. doi: 10.3748/wjg.v11.i16.2513. PMID 15832428
- [Result] Dery L, Galambos Z, Kupcsulik P, Lukovich P. [Cirrhosis and cholelithiasis. Laparoscopic or open cholecystectomy?]. Orv Hetil. 2008 Nov 9;149(45):2129-34. doi: 10.1556/OH.2008.28450. Hungarian. PMID 18977740
- [Result] Vu T, Aguilo R, Marshall NC. Clipless technique of laparoscopic cholecystectomy using the harmonic scalpel. Ann R Coll Surg Engl. 2008 Oct;90(7):612. doi: 10.1308/rcsann.2008.90.7.612a. No abstract available. PMID 18831871
- [Result] Bessa SS, Al-Fayoumi TA, Katri KM, Awad AT. Clipless laparoscopic cholecystectomy by ultrasonic dissection. J Laparoendosc Adv Surg Tech A. 2008 Aug;18(4):593-8. doi: 10.1089/lap.2007.0227. PMID 18721011
- See also: Mansoura University Hospital — http://home.mans.eun.eg